CLINICAL TRIAL: NCT00244179
Title: New Immunomodulatory Therapy Strategies in Chronic Reactive Arthritis: Immunostimulation Plus Antibiotic Versus Immunosuppression Plus Antibiotic Versus Conventional Standardtherapy
Brief Title: New Immunomodulatory Therapy Strategies in Chronic Reactive Arthritis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: dfg (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: ReA01
Record Dates: First submitted 2005-10-24; First posted 2005-10-26 (Estimated); Last update posted 2006-09-08 (Estimated); Status verified 2006-09

CONDITIONS: Reactive Arthritis
Keywords: reactive arthritis; trial; interferon-gamma; infliximab; chronic; tnf-blocker
MeSH Terms: conditions — Arthritis, Reactive; Bronchiolitis Obliterans Syndrome | interventions — Interferon-gamma; Infliximab; Antirheumatic Agents

INTERVENTIONS:
Drug: interferon-gamma
Drug: infliximab
Drug: dmard

SUMMARY:
1. to investigate, whether one of the two alternative therapy strategies (antibiotic plus immunostimulation versus antibiotic plus immunosuppression) in chronic reactive arthritis is therapeutical superior to conventionel standardtherapy (DMARD).
2. to investigate, whether one or more of the different therapy strategies cause an altered detection of bacterial DNA in the joint or colon.
3. to measure the antigen-specific and -unspecific immune response (predominantly t-cell response) during therapy and correlate it with the clinical course.
4. to gain knowledge from these analyses and the clinical course concerning the pathogenesis and the point of attack for possible therapies in chronic reactive arthritis.
5. to compare cytokine-profiles of CD4- and CD8-positive T-cells from patients treated with infliximab to those treated with etanercept.

DETAILED DESCRIPTION:
Studybackground Enteric reactive arthritis (ReA) is an extraintestinal manifestation of an infection of colon mucosa caused by enterobacteria. At least in the chronic courses of ReA a bacterial persistence can be assumed which is most likely to be located in colon mucosa or colon associated lymph nodes. The persistence of bacteria might be in consequence of an insufficient t-helper-immune-response.

On the other hand the persistence of the pathogen itself could be harmless and the local immune-pathology could be caused by a hypersensitivity immune response The project in hand shall assess whether 1.) immune stimulation or immune suppression is the best therapy for chronic reactive arthritis and 2.) enteric reactive arthritis is based on bacterial persistence or a hypersensitivity immune response.

By gaining these data we hope to be able to draw conclusions concerning the pathogenesis and therapies of other infections that affect the mucosa.

ReA occurs after infection of the intestine (enteric ReA) or after urogenital infection caused by chlamydia (urogenital ReA). Both forms of ReA are pathogenetically und immunogenically closely related and are treated as one entity.

Patients who are enrolled in the trial with enteric ReA (colon as possible location of bacterial persistence), not those with urogenital ReA (location of bacterial persistence not known) undergo colonoscopy before and after treatment-period to obtain colon biopsies for further work up.

Patients with knee involvement (arthritis of knee) undergo arthroscopy before and after treatment-period to obtain synovial biopsies for further work up.

Recently collected data form our group concerning patients with ankylosing spondylitis under therapy with infliximab or etanercept have shown that the potential of CD4- and CD8-positive t-cells to produce interferon gamma (IFN Gamma) or tumornecrosisfactor alpha (TNF-Alpha) after antigen-specific or -unspecific stimulation was distinct reduced under therapy with infliximab, whereas this potential under therapy with etanercept increased.

In context with recently collected data concerning Crohn´s disease it can be assumed that by binding not only soluble TNF-Alpha but as well membrane-associated TNF-Alpha infliximab induces apoptosis of t-cells, whereas etanercept induces no apoptosis. These results could explain, why infliximab but not etanercept is effective in treating Crohn´s disease Furthermore the induction of apoptosis could explain why therapy with infliximab is associated with a higher incidence of tuberculosis compared to etanercept.

By means of FACS (Fluorescence activated cell sorting) we want to examine, whether TNF-blocking agents in patients with chronic ReA induce a t-cell-suppression and compare the cytokine-pattern of CD4- and CD8-positive t-cells from patients treated with infliximab with the cytokine-pattern of CD4- and CD8-positive t-cells from patients treated with etanercept.

The comparison of both therapies - infliximab and etanercept - is of special interest, because both TNF-blocking agents obviously have a different active profile as well as different side effects.

Background for dosage Ciprofloxacin 2 x 500 mg p.o. daily is conventional therapy for treating infections with enterobacteria.

Clinical trials with infliximab 5 mg/kg in patients suffering from ankylosing spondylitis have been successfully performed. Dosages of infliximab 1 - 10 mg/kg have been used in treating succesfully patients with rheumatoid arthritis. A dosage of 5 mg/kg was more effective than 1 mg/kg, but 10 mg/kg was only slightly better. Infliximab has been approved for the indication rheumatoid arthritis and ankylosing spondylitis.

Clinical trials with etanercept 25 mg s.c. 2 x per week in patients suffering from ankylosing spondylitis and rheumatoid arthritis have been performed successfully and effectively. Etanercept has been approved for the indication ankylosing spondylitis, rheumatoid arthritis and psoriasic-arthritis.

To treat patients suffering from tuberculosis who do not respond to conventional anti-tuberculosis-therapy IFN-g (interferon-gamma) 3 x 100 - 150 µg/week s.c. has been succesfully administered.

In a clinical trial to assess the efficacy in rheumatoid arthritis IFN-g 50 µg was administered daily during the first three weeks and every other day in the last week.

Patients who receive standard-therapy (Sulphasalazine, Methotrexate, Leflunomide) are treated with common dosages of these drugs that are deduced from the common treatment of rheumatoid arthritis.

Background for selection of patients 80% of patients suffering from acute ReA heal up within 6 months. About 40% of patients have severe symptoms for more than 6 months and about 20% develop a chronic course of arthritis.

These patients with chronic ReA are regrettably insufficiently treated with the available drugs (NSAID, Methotrexate, Sulphasalazine, Leflunomide).

Patients who are enrolled in this trial have to have a definite chronic ReA (disease duration of at least 12 months), a joint pain of > 4 (visual analogue scale, 0-10), a constant demand of NSAID and an active arthritis affecting at least one joint.

ELIGIBILITY:
Inclusion Criteria:

1. definite classification of the arthritis as ReA enteric ReA is defined as an arthritis, which occurs within 4 weeks after a preceding symptomatic infection of the gut with enteric bacteria such as yersinia, salmonella, campylobacter jejuni, shigella. If no symptomatic preceding infection can be remembered the triggering enterobacterium has to be clearly identified by serology or stool culture. Other causes for a diarrhea like for example inflammatory bowel disease have to be eliminated.

   urogenital (chlamydia-triggered) ReA is defined as an arthritis, which occurs within 4 weeks after a symptomatic urogenital infection or an infection of the upper airways or if chlamydia can be clearly identified be serology or direct proof.
2. disease duration > 12 months
3. age 18 to 70 years
4. active arthritis in at least one joint
5. constant demand of NSAIDs
6. intensity of pain > 4 on a visual analogue scale (VAS; 0 to 10)
7. patients are allowed to have been treated with so-called conventional therapy (Sulphasalazine, Methotrexate etc.) or steroids i.a. before, but they have to be stopped 4 weeks before enrolled into the trial
8. able to self-administer s.c. injections or have a caregiver who will do so
9. women of child bearing potential must have a negative pregnancy test at study baseline and use an adequate, effective method of contraception (such as implants, injectables, combined oral contraceptives, some IUDs, sexual abstinence, vasectomised partner) for a duration of 6 months after stop of therapy. Sexual active men must use an accepted method of contraception for a duration of 6 months after stop of therapy.
10. reading a normal chest/ lung x-ray, negative Mendel-Mantoux-skin test (10,0 TE) (both not older than 4 weeks). If Mendel-Mantoux-skin test is positive and / or there are hints for a healed up tuberculosis in the chest x-ray (latent tuberculosis) and the patient shall receive infliximab or etanercept an additional therapy with isoniazid 300 mg daily starting 4 weeks before first administration of infliximab or etanercept has to be given.
11. signed informed consent

Exclusion Criteria:

1. female subjects who are pregnant or breast-feeding
2. previous treatment with cytokines or anti-cytokines (biological agents)
3. severe infections within the last 3 months
4. history of opportunistic infections within the last 2 months (herpes zoster, cytomegaly virus-, pneumocystis carinii-infection)
5. HIV-infection
6. history of malignancy
7. receipt of any live (attenuated) vaccines within last 30 days before screening visit
8. previous diagnosis or signs of demyelinating diseases
9. history of uncontrolled diabetes, unstable ischemic heart disease, active inflammatory bowel disease, active peptic ulcer disease, recent stroke, ongoing congestive heart failure, and any other condition which, in the opinion of the investigator, would put the subject at risk by participation in the protocol.
10. history of cytopenia
11. laboratory exclusions are: hemoglobin level < 8,5 g/dl, white blood cell count < 3.5 x109/l, platelet count < 125 x 109 /l, creatinine level > 175 µmol/ liver enzymes > 1,5, alkaline phosphatase >2 times the upper limit of normal, Quick > 50.
12. clinical examination showing significant abnormalities of clinical relevance
13. participation in trials of other investigational medications within 30 days of entering the study
14. history or current evidence of abuse of "hard" drugs (e.g. cocaine/heroine)
15. current medication with 7,5 mg or more Prednisolon daily

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2003-01

PRIMARY OUTCOMES:
change in intensity of pain (VAS pain, scale 0-10)
change in funcion (WOMAC)

SECONDARY OUTCOMES:
decrease of CRP/ESR
change of cytokine response
change of DNA detection
number of swollen and tender joints
number of entheseal localisations
improvement of quality of life, "Short form 36" (SF-36)
BASDAI (disease activity index)
Reduction of NSAIDs
Patient's global (scale 0-10).
Physician's global (scale 0-10).

CONTACTS AND LOCATIONS:
Overall Officials: joachim sieper, prof., Principal Investigator — charite, campus benjamin franklin, rheumatology, berlin
Locations (1):
- Charite Campus Benjamin Franklin, Rheumatology, Berlin, Germany